CLINICAL TRIAL: NCT05903482
Title: Gastric Volume in Patients on GLP-1 Medications
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 23-021125
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetic, in GLP-1 RA: non-invasive, gastric ultrasound in children who are on GLP-1 RA medications and have type 2 diabetes mellitis (DM) and/or obesity and/or type 1 DM
  Interventions: Other: None - observational
- Diabetic, not on GLP-1 RA: non-invasive, gastric ultrasound in children who are not on GLP-1 RA medications and have type 2 diabetes mellitis (DM) and/or obesity and/or type 1 DM.
  Interventions: Other: None - observational
- Non-diabetic, not on GLP-1 RA: non-invasive, gastric ultrasound in non-diabetic children who are not on GLP-1 RA medications and do not have diabetes or obesity.
  Interventions: Other: None - observational

INTERVENTIONS:
Other: None - observational — Observational

SUMMARY:
Evaluating gastric volume in patients on GLP-1 RA medications

DETAILED DESCRIPTION:
Glucagon like peptide 1 (GLP-1) receptor agonist (RA) medications have in recent years been approved for use in children with type 2 diabetes mellitis (DM) and obesity. The side effects of these medications include nausea and vomiting, and in the adult literature, delayed gastric emptying has been described. Due to the likelihood of delayed enteric motility, standard nil per os (NPO) guidelines may not be sufficient to minimize the chance of aspiration of gastric contents before anesthesia and surgery in patients receiving GLP-1 RA medications.

Investigators seek to measure the gastric volume of children on GLP-1 RA medications who are appropriately NPO (greater than/equal to 8 hours for solids and greater than/equal to 1 hour for clear liquids) using standard institutional NPO guidelines. The secondary objective is to measure the gastric volume of children not on GLP-1 RA medications, but with type 2 diabetes mellitis or obesity and/or type 1 DM.

The only study intervention is the addition of a gastric ultrasound. The gastric ultrasound is a non-invasive mode of imaging using sound waves with no known safety risks. The ultrasound will be performed while the subject is awake and will take less than 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

Fasting Diabetic On GLP-1 RA

Exclusion Criteria:

Prior surgery that affects gastric anatomy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Fasting children on GLP-1 RA
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Gastric volume in pediatric patients on GLP-1 RA | Day 1
  A non-invasive, ultrasound will be performed to assess gastric volume. A second investigator not performing the ultrasound and blinded to whether the subject is taking a GLP-1 RA medication and whether the patient has diabetes and/or obesity will then assess the ultrasound images qualitatively for gastric contents (empty, clear liquids, solids) and quantitatively for gastric fluid volume if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Elaina Lin, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No